CLINICAL TRIAL: NCT04782765
Title: Phase Ⅱ Trial of Neoadjuvant Chemotherapy Combined With Camrelizumab Followed by Chemoradiotherapy in Patients Without Distant Metastasis Nasopharyngeal Carcinoma
Brief Title: Phase Ⅱ Trial of Camrelizumab in Patients Without Distant Metastasis Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Peiguo Wang, Chief Physician, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-TJ-CC-HNC-II-002
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Disease-free Survival Rate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Chemotherapy+Chemoradiotherapy (Experimental): Patients received neoadjuvant Camrelizumab 200mg combined with chemotherapy (Cisplatin 20mg/m2, Day 1-3, Docetaxel 75mg/m2, Day 1) for 2 cycles every 21 days, followed by concurrent chemoradiotherapy with Camrelizumab monotherapy maintenance
  Interventions: Drug: Camrelizumab+Chemotherapy+Chemoradiotherapy

INTERVENTIONS:
Drug: Camrelizumab+Chemotherapy+Chemoradiotherapy — Patients received neoadjuvant Camrelizumab 200mg combined with chemotherapy (Cisplatin 20mg/m2, Day 1-3, Docetaxel 75mg/m2, Day 1) for 2 cycles every 21 days, followed by concurrent chemoradiotherapy with Camrelizumab monotherapy maintenance

SUMMARY:
To see the effect if a combination of neoadjuvant chemotherapy combined with Camrelizumab followed by chemoradiotherapy in treating patients without distant metastasis nasopharyngeal carcinoma

DETAILED DESCRIPTION:
The primary objective of this phase 2 study is to assess disease-free survival rate of 3 years in patients with NPC. The secondary objective is to observe objective response rate, progression free survival, overall survival and safety

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent before enrollment;
* Male or female under the age of 70;
* Diagnosed by imaging examination and histopathologic examination Ⅱ I - Ⅳ b period in patients with nasopharyngeal carcinoma
* No first-line treatment has been received
* ECOG/PS score: 0 ~ 1;
* Expected survival is greater than 12 weeks;
* The function of vital organs meets the following requirements (excluding the use of any blood components and cell growth factors within 14 days) :

  1. Routine blood examination (no blood transfusion or use of hematopoietic stimulant subclass drugs to correct within 14 days before screening) Hemoglobin (Hb) ≥90 g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Absolute value of lymphocyte count (LC) ≥0.5×109/L; Platelet count (PLT) ≥100×109/L; White blood cell count (WBC) ≥4.0×109/L and ≤15×109/L;
  2. Biochemistry (no blood transfusion or albumin within 14 days prior to screening) AST and ALT ≤2.5 x ULN ALP ≤ 2.5 x ULN TBiL≤ 1.5 x ULN ALB≥30 g/L; Cr≤1.5×ULN, and creatinine clearance rate (CrCl)≥80 mL/min (Cockcroft-Gault formula)
* Normal coagulation function, no active bleeding and thrombotic disease A. International standardized ratio INR≤1.5×ULN; B. Partial thromboplastin time APTT≤1.5×ULN; C. Prothrombin time Pt ≤1.5×ULN;
* For women of non-surgical sterilization or reproductive age, use of a medically approved contraceptive method (such as intrauterine device, birth control pills or condoms) during the study treatment period and within 3 months after the end of the study treatment period;Women of reproductive age who are not surgically sterilized must be negative for serum or urine HCG within 7 days prior to study enrolment;And must be non-lactation;Male patients who are not surgically sterilized or of reproductive age need to agree to use a medically approved method of contraception with their spouse for the duration of the study treatment period and for three months after the end of the study treatment period.
* Subjects volunteered to participate in this study, with good compliance, safety and survival follow-up.

Exclusion Criteria:

* Previous radiation, chemotherapy, hormone therapy, surgery, or molecular targeted therapy;
* Imaging confirmed patients with distant metastasis;
* Subjects have previous or co-existing malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* Previous treatment with carrelizumab or other PD-1/PD-L1 inhibitors was not included;Subject is known to have a prior allergy to macromolecular protein formulations or to any of the carrizumab or chemotherapy ingredients used by the subject during neoadjuvant therapy;
* there is no active participants autoimmune disease or a history of autoimmune diseases (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, the pituitary gland inflammation, vasculitis, nephritis, thyroid function, thyroid function is reduced, always had thyroid surgery must be incorporated into;Subjects with vitiligo or asthma that had been in complete remission during childhood were enrolled as adults without any intervention;Asthmatic subjects requiring bronchodilators for medical intervention were not included);
* Subjects are using immunosuppressants and continue to use them within 2 weeks before enrolment;
* Patients with clinical cardiac symptoms or diseases that are not well controlled, such as :(1) NYHA2 heart failure or above, (2) unstable angina, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
* Abnormal coagulation function (PT>16 s, APTT>43S, TT>21 s, Fbg>2g/L) with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
* Previous or current severe bleeding (bleeding within 3 months >30 ml), hemoptysis (within 4 weeks >5 ml fresh blood) or thromboembolic events (including stroke events and/or transient ischemic attack) within 12 months;
* Subjects were still using TCM immunomodulator 2 weeks before enrollment;
* Subjects have active infection or unexplained fever during screening or prior to first administration >38.5 degrees (subject fever due to tumor can be included, as determined by the investigator);
* Patients with previous and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe pulmonary function impairment, etc.;Subjects who still had grade ≥2 peripheral neuropathy within 3 days before the first medication;
* Subjects with congenital or acquired immune deficiency, such as HIV infection, or active hepatitis (transaminase does not meet the inclusion criteria, hepatitis B reference: HBV DNA≥1000 IU/ml;Reference for hepatitis C: HCV RNA≥1000 IU/ml); Chronic hepatitis B virus carriers with HBV DNA < 2000 IU/ mL must receive antiviral therapy during the trial to be enrolled.
* Live vaccine was administered less than 4 weeks before or possibly during the study period;
* Subject has a known history of psychotropic substance abuse, alcohol abuse or drug abuse;
* Subjects received traditional Chinese medicine treatment within 4 weeks before the first treatment;
* Subject is unable or does not agree to bear the cost of examination and treatment at their own expense, except for clinical investigational drugs, combined chemotherapy and SAE related to clinical investigational drugs combined chemotherapy;
* Researchers think that should be left out in this study, the researchers determine, for example, the subjects have other factors that may result in this study were forced to midway termination, such as, other serious disease (including mental illness) need to merge treatment, there are serious abnormal laboratory examination, accompanied by factors such as family or society, will affect the safety of the subjects, or information and the collection of the sample.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2021-03-20 (Estimated); Primary Completion 2023-03-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival（DFS）rate of 3 years | 3 years
  Disease-free survival is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Overall response rate | 16 weeks after completion of concurrent chemoradiotherapy
  Tumour response was classified according to RECIST, version 1.1
Distant metastasis-free survival(DMFS) rate of 3 years | 3 years
  The DMFS rate is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Incidence of adverse events | 3 years
  Incidence of adverse events is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE)5.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme

CONTACTS AND LOCATIONS:
Locations (1):
- Peiguo Wang, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Wang Z, Sun Y, Wang Q, Chai Y, Sun J, Zhang X, Wang Q, Wang W, Wang P. Induction chemotherapy plus camrelizumab combined with concurrent chemoradiotherapy in locoregionally advanced nasopharyngeal carcinoma in non-endemic areas: a phase 2 clinical trial in North China. BMC Med. 2025 Feb 27;23(1):126. doi: 10.1186/s12916-025-03964-9. PMID 40016735